CLINICAL TRIAL: NCT02735967
Title: The Use of Diadynamic in Association With a Manual Therapy Program for Patients With Impingement Syndrome: a Randomized Blind Clinical Trial
Brief Title: The Use of Diadynamic in Association With a Manual Therapy Program for Patients With Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Cid André Fidelis de Paula Gomes, Phd, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 50917515.3.0000.5511
Record Dates: First submitted 2016-04-02; First posted 2016-04-13 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Shoulder Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group manual therapy + diadynamic (Experimental): Initially, the positional release techniques will be performed while maintaining this position for 90 seconds procedure is repeated 3 times. Then, the therapist performs the ischemic compression technique on the myofascial trigger point, the compression is maintained for 90 seconds by 3 replications.
  Through an electrotherapy device were applied diadynamic in that myofascial trigger point previously marked. 4 minutes from the fixed two-phase mode will be applied (DF), 4 minutes long periods (LP) and 4 minutes short periods (CP), the first and second intensely in the sensitive line and the third motor threshold, both supportable according to each patient.
  Interventions: Other: manual therapy; Device: diadynamic current
- Group manual therapy (Active Comparator): Initially, the positional release techniques will be performed while maintaining this position for 90 seconds procedure is repeated 3 times. Then, the therapist performs the ischemic compression technique on the myofascial trigger point, the compression is maintained for 90 seconds by 3 replications.
  Interventions: Other: manual therapy
- Group diadynamic (Active Comparator): An electrotherapy device were applied diadynamic in that myofascial trigger point previously marked. 4 minutes from the fixed two-phase mode will be applied (DF),4 minutes long periods (LP) and 4 minutes short periods (CP), the first and second intensely in the sensitive line and the third motor threshold, both supportable according to each patient.
  Interventions: Device: diadynamic current

INTERVENTIONS:
Other: manual therapy — the positional release techniques will be performed while maintaining this position for 90 seconds procedure is repeated 3 times. Then, the therapist performs the ischemic compression technique on the myofascial trigger point, the compression is maintained for 90 seconds by 3 replications.
  Arms: Group manual therapy; Group manual therapy + diadynamic
Device: diadynamic current — Through an electrotherapy device were applied diadynamic in that myofascial trigger point previously marked. 4 minutes from the fixed two-phase mode will be applied (DF), 4 minutes long periods (LP) and 4 minute short periods (CP), the first and second intensely in the sensitive line and the third motor threshold, both supportable according to each patient.
  Arms: Group diadynamic; Group manual therapy + diadynamic

SUMMARY:
The aim of this study will be to evaluate the effects of the use of manual therapy and diadynamic in muscle trigger points in the upper trapezius muscle in individuals diagnosed with shoulder impingement syndrome, unilateral shoulder as functional capacity, pain intensity and pain threshold the pressure.

ELIGIBILITY:
Inclusion Criteria:

* history of anterior lateral and unilateral shoulder pain
* with more than 3 months duration
* intensity of at least 4 points on the Numerical Rating Pain Scale
* positivity in at least 2 of 3 orthopedic tests for impingement syndrome: Neer, Hawkins or Jobe
* Associated with these characteristics volunteers should submit myofascial trigger points unilateral and active, centrally located in the trapezius muscle descending fibers associated with painful shoulder

Exclusion Criteria:

* diagnosis of bilateral impingement syndrome shoulder
* fibromyalgia
* muscle injury
* history of trauma on the shoulder
* ruptured tendons
* ligamentous laxity
* symptoms of numbness and / or tingling in the upper limbs
* corticosteroid injection use shoulder
* making use of anti-inflammatory
* they performed surgery or physical therapy treatment in the last 6 months in the affected shoulder.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
shoulder disability | Change from Baseline in the Shoulder Pain and Disability Index at 4 weeks
  questionnaire of quality of life developed to assess pain and associated with specific inability to shoulder disorders.

SECONDARY OUTCOMES:
intensity of pain | Change from Baseline in The Numerical rating pain scale at 4 weeks
  the Numerical rating pain scale, a simple, easily administered scale evaluates
level of pressure pain | change from Baseline in ThePressure Pain Threshold at 4 weeks
  Pressure Pain Threshold in the shoulder with algometer dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Cid André Fidelis de Paula Gomes, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Related Info — http://www.uninove.br